



"2021, Año de la Independencia"

| | Ciudad de México, a | de | de 2020. |
|---|---|---|---|
| CONSENTIMIENTO INFORMADO - Título del protocolo: Nuevo régimen de PROFILAXIS | | | |
| para infección por SARS-CoV-2 en profesionales de la salud con dosis bajas de Hidroxicloroquina | | | |
| y Bromhexina. Un ensayo clínico aleatorizado doble ciego placebo control (ELEVATE Trial). | | | |
| Nombre del investigador principal/coordinador: Dr. Julio Granados Montiel | | | |
| Nombre del sujeto de investigación: | | | |
| | <u> </u> | | |

A través de este documento, que forma parte del proceso para la obtención del consentimiento informado, me gustaría invitarlo a participar en la investigación titulada: "Nuevo régimen de PROFILAXIS para infección por SARS-CoV-2 en profesionales de la salud con dosis bajas de Hidroxicloroquina y Bromhexina. Un ensayo clínico aleatorizado doble ciego placebo control (ELEVATE Trial)". Antes de decidir, necesita entender por qué se está realizando esta investigación y en qué consistirá su participación. Por favor tómese el tiempo que usted necesite para leer la siguiente información cuidadosamente. Puede enviarnos un correo electrónico a profilaxiscovid@gmail.com para contestar tus dudas y preguntas acerca de esta investigación.

- 1. ¿Dónde se llevará a cabo esta investigación? Esta investigación se llevará a cabo en el Instituto Nacional de Rehabilitación, situado en la zona de hospitales de la Alcaldía Tlalpan.
- **2.** ¿Cuál es el objetivo de esta investigación? El objetivo de nuestra investigación es valorar la eficacia del uso de Hidroxicloroquina combinado con Bromhexina en personal de salud sano y expuesto a la atención de pacientes con sospecha o confirmación de SARS-CoV-2, para prevenir la infección por este virus. Esta prevención es una profilaxis; significa la protección antes de desarrollar un padecimiento tomando alguna medida, en el caso de esta investigación será con las medicinas antes mencionadas.
- 3. ¿Por qué es importante esta investigación? Esta investigación es importante porque busca determinar si es posible prevenir que el personal que labora en hospitales y está en riesgo de contagio por el virus SARS-CoV2 ("nuevo coronavirus") desarrolle la enfermedad COVID-19, mediante una combinación de los medicamentos hidroxicloroquina (HCQ) y bromhexina (BHX). La labor de los profesionales de la salud es esencial, por lo que es fundamental evitar que se enfermen, ya que están en un riesgo constante, peor aún que se puedan requerir de hospitalización para curarse o hasta perder la vida. Se calcula que, en Italia, el 20% del total de los trabajadores de la salud fueron contagiados por coronavirus.
- **4.** ¿Por qué he sido invitado a participar en esta investigación? Le invitamos a participar en esta investigación del Instituto Nacional de Rehabilitación para buscar un tratamiento preventivo para la infección por SARS-CoV-2 en personal de salud expuesto, por ser un profesionista en primera línea de atención de pacientes con sospecha o confirmación de la infección: médicos, enfermeras, camilleros, técnicos en urgencias médicas, técnicos de rayos X y de laboratorio. Los criterios de inclusión para participar son:

Calzada México Xochimilco No. 289 Col. Arenal de Guadalupe, Alcaldía Tlalpan Ciudad de México., C.P. 14389 Tel. (55) 5999 1000 ext. 19610 y 19604





"2021, Año de la Independencia"

- Laborar en hospitales públicos de cualquier sistema u hospital privado que atiende a pacientes con sospecha o confirmación de enfermedad COVID-19.
- Edad mayor de 18 años y menor de 60 años,
- Sexo masculino o femenino
- Expuesto a la atención de pacientes con sospecha o confirmación de infección por SARS-CoV-2.
- **5. ¿Estoy obligado a participar?** Su participación es voluntaria, anónima y confidencial; no tiene que participar forzosamente. No habrá impacto negativo alguno si decide no participar en la investigación, y no demeritará de ninguna manera la calidad de la atención que reciba en el Instituto Nacional de Rehabilitación "Luis Guillermo Ibarra Ibarra", en término de sus derechos como paciente, o en caso de ser empleado de esta institución, sus derechos como trabajador.
- **6.** ¿En qué consiste mi participación y cuánto durará? Si usted decide participar en esta investigación, seguirá el proceso de reclutamiento que consiste en 3 fases, en *2 citas* en el INR. Se realizará una historia y análisis clínicos iniciales, que incluirá la toma de un hisopado de secreciones nasofaríngeas para la prueba molecular de reacción en cadena de polimerasa con transcriptasa reversa (RT-PCR, por sus siglas en inglés) que detecta la presencia del virus SARS-CoV-2 y de 30 mililitros de sangre de una vena periférica para biometría hemática, química sanguínea y determinación de anticuerpos (Inmunoglobulinas G y M) contra el mismo virus. Adicionalmente se realizará un electrocardiograma (EKG) y un examen de fondo de ojo.

La primera cita es para hacer el hisopado de secreciones nasofaríngeas para la RT-PCR. Este procedimiento es poco molesto y es rápido, y dura 10 minutos aproximadamente. Se realiza en un área especializada. Usted será recibido/a en la entrada del hospital previa cita temprano en la mañana, donde la acompañará uno de los médicos del protocolo. Después de la toma del hisopado podrá retirarse.

Si la prueba sale POSITIVA, se le recomendarán medidas de manejo por parte de un infectólogo para cuidarse. No proseguirá con la siguiente etapa de evaluación para el estudio. Si saliera NEGATIVA para la 'presencia del virus SARS-CoV-2, entonces proseguirá con la siguiente fase de evaluación.

Posteriormente, se le realizará una breve historia clínica y se le tomarán muestras de sangre para laboratorio y se realizarán tanto el EKG como el examen de fondo de ojo. Debe prever aproximadamente 3 horas de su día, entre las 8h00 AM y 11h00 AM, y NO MANEJAR ya que la dilatación de la pupila necesaria para el fondo de ojo causa visión borrosa por 6 a 8 horas. Previa cita será recibido por un médico del protocolo, y la historia clínica, toma de sangre para laboratorio y EKG serán realizados en el servicio de Urgencias del INR. Posteriormente será llevado al área de Oftalmología donde se le colocarán unas gotas para dilatar la pupila. El efecto puede tardar hasta 30 minutos para hacer efecto, después de lo cual se realiza el examen del fondo de ojo y análisis de la pupila para discernir cualquier anomalía. Posterior al examen podrá retirarse.

La finalidad del EKG es establecer si Ud. tiene alguna arritmia cardíaca, y el fondo de ojo para determinar si hay cambios a nivel de la retina. Se han descrito efectos adversos con el uso a largo plazo de la HCQ: lesiones maculares en retina (2% a 10 años de dosis cumulativa) y alargamiento del intervalo QT que clínicamente no tiene repercusiones pero en asociaciones con otres.





"2021, Año de la Independencia"

medicamentos puede causar trastornos del ritmo cardíaco. Por lo anterior, en caso de detectarse una anomalía en su retina o EKG, no podrá participar en el estudio.

Si su examen de sangre revela la presencia de inmunoglobulinas M o G (IgM/G) contra el virus del COVID-19, usted no necesitará participar en el estudio: Ya estuvo expuesto y tiene inmunidad contra la enfermedad.

Si sus pruebas RT-PCR y IgM/G son negativas y no presenta anomalías en su EKG ni en el examen de fondo de ojo, podrá participar en esta investigación. Se le asignará a uno de dos grupos: recibe medicamento (experimental) o recibe placebo (control).

Esta asignación de en qué grupo estará será mediante un programa de computadora y totalmente al azar. Ni los investigadores ni Usted sabrán en ningún momento, a que grupo fue asignado. De ser asignado al grupo de experimental o intervención, recibirá los 2 medicamentos comerciales con su fórmula activa: Hidroxicloroquina 200 miligramos una vez al día y Bromhexina 8 miligramos cada 8 horas. Si usted fuera asignado al grupo control o placebo, recibirá dos pastillas que simulan cada una la presentación comercial de los medicamentos del grupo experimental pero sin el principio activo o fármaco (placebo). El propósito de tener un grupo control es para evaluar el verdadero efecto del tratamiento con la combinación de los medicamentos Hidroxicloroquina y Bromhexina.

El tratamiento (medicamento o placebo) se le entregará al firmar el presente consentimiento informado para participar en esta investigación, en el servicio de Vigilancia Epidemiológica del Instituto; se le proporcionará el tratamiento para 30 días inicialmente, al término de los cuales se realizará la 1ª evaluación clínica y se le entregará entonces tratamiento para completar los 60 días cuando se realizará la evaluación final que concluye su participación en el estudio.

Durante la investigación, se evaluará semanalmente por vía telefónica o correo electrónico cualquier posible evento adverso, reacción secundaria, síntomas de COVID-19 y la adherencia al tratamiento.

A los 30 y 60 días de haber iniciado su participación, se realizará una evaluación clínica que incluye un pequeño cuestionario, toma de signos vitales repetir el hisopado y toma de sangre para las pruebas diagnósticas de RT-PCR y determinación de IgM/IgG. En la evaluación final a los 60 días se tomará además un nuevo EKG y otro examen de fondo de ojo con dilatación de pupilas. Si usted resulta positivo en cualquiera de las 2 pruebas para COVID-19 durante la evaluación 30 días se le dará de baja del estudio, pero seguirá siendo monitoreado hasta los 60 días.

El siguiente diagrama de flujo muestra los pasos a seguir desde que usted ha sido invitado a participar:







geniería de Tejidos Terapia r y Medicina Regenerativa









"2021, Año de la Independencia"

- 7. ¿Cuáles son los beneficios de formar parte de esta investigación? Las ventajas de participar a esta investigación es de conocer si está o ha estado infectado por el SARS-CoV-2 durante las 3 evaluaciones clínicas además de conocer si tiene o no alteraciones en retina y corazón. Esto le permite tomar decisiones médicas, y en el caso de ser portador poder tomar medidas con sus familiares. Adicionalmente estará participando en un estudio que contribuye al conocimiento sobre la eficacia de un tratamiento para proteger al personal sanitario expuesto al virus SARS-CoV-2.
- **8.** ¿Existe alguna alternativa que pueda proporcionarme mayor beneficio que lo que me proponen en esta investigación? No; hoy en día no existe ningún medicamento o alternativa farmacológica que esté probado para brindar un mayor beneficio o protección contra esta enfermedad. El uso correcto del Equipo de Protección Personal, y las recomendaciones de distanciamiento social y evitar tocarse la cara y el lavado frecuente de manos son por ahora las únicas medidas de protección eficaz.
- 9. ¿Cuáles son los posibles riesgos de formar parte de esta investigación? Los posibles riesgos, en caso de ser asignado al grupo de intervención, son las reacciones adversas reportadas en la literatura de los 2 medicamentos que investigamos. Estas reacciones se han reportado en menos del 5% de los pacientes con tratamientos de mayor dosis o y tiempos de administración de varios años que los prescritos por 60 días de esta investigación; sin embargo, no se descarta que usted pudiera tener alguno de estos efectos adversos. Los efectos adversos reportados son:
- Alteraciones del corazón y vasos sanguíneos como alteraciones en el músculo del corazón, alteraciones de la conducción eléctrica en el corazón (arritmias), así como crecimiento del corazón.
- Alteraciones del hígado como anormalidades de la función o inflamación del hígado.
- Alteraciones gastrointestinales como diarrea, perdida de hambre, náusea, dolor abdominal y, en raras ocasiones, vómito.
- Alteraciones sanguíneas como anemia (baja producción de glóbulos rojos) o leucopenia (disminución de la producción de glóbulos blancos).
- Alteraciones del metabolismo y nutrición como hipoglucemias (baja de la concentración de glucosa en sangre).
- Alteraciones neuromusculares como miopatía esquelética o neuromiopatía, debilidad progresiva y atrofia muscular.
- Alteraciones del sistema inmune como urticaria, angioedema y broncoespasmo.
- Alteraciones de los ojos, como alteraciones en la retina con cambios en la pigmentación y
  defectos en el campo visual, visión anormal del color, cambios en la córnea, visión borrosa,
  sensibilidad a la luz.
- Alteraciones en la piel como ampollas, descamación, enrojecimiento, comezón, aumento en el número de canas y caída de cabello. Si usted padece de psoriasis, este será un criterio de exclusión.
- Alteraciones neuro-psiquiátricas como dolor de cabeza, convulsiones, temblor, nerviosismo, fragilidad emocional, sentir que otros te están mirando o controlando tu comportamiento, que otros pueden escuchar tus pensamientos, ver u oír cosas que no están allí, o comportamiento suicida.
- Alteraciones auditivas o del equilibrio como mareo, zumbido de oídos, percepción de ruidos, disminución de la capacidad auditiva.





"2021, Año de la Independencia"

- 10. ¿Tendré alguna molestia durante y/o después de mi participación? Usted podría presentar molestias durante su participación en el momento de la toma de muestras sanguíneas (punción venosa) así como en la toma de las muestras de hisopado nasofaríngeo. Las molestias a causa de los medicamentos tomados podrían ser por la presencia de efectos adversos de los mismos (descritos arriba). Con relación a después de su participación, estudios publicados demuestran que pacientes que han tomado esta dosis durante 60 días, tienen el medicamento en sangre durante los 120 días subsecuentes, desapareciendo totalmente las molestias que se hayan podido presentar al terminar este periodo.
- 11. ¿Recibiré alguna compensación por mi participación? Usted no recibirá ninguna compensación económica o de otra naturaleza por su participación en esta investigación.
- **12. ¿Tendrá algún costo para mí, participar en esta investigación?** Para usted NO tendrá costo alguno la participación, los medicamentos, consultas médicas, los estudios de laboratorio y gabinete (3 hisopados y toma de sangre para pruebas diagnósticas, 2 electrocardiogramas y 2 exámenes de fondo de ojo) serán totalmente gratuitos.
- 13. Una vez que acepte mi participación, ¿es posible retirarme de la investigación? Usted podrá retirarse de la investigación en todo momento, sin tener que otorgar ninguna explicación para lo mismo.
- 14. ¿En qué casos se me puede suspender de la investigación? A usted se le puede suspender de la investigación inmediatamente si llegara a presentar algún efecto colateral de los medicamentos descritos en el punto 9 que pongan en riesgo su salud y/o su vida, y usted recibirá la atención medica necesaria para revertir, de ser posible, estos efectos colaterales sin costo alguno. Podría presentarse una reacción de hipersensibilidad (alergia) a alguno de los medicamentos, y las alteraciones del ritmo cardíaco o de retina se presentan rara vez pero después de años de dosis cumulada entonces es poco probable que se presente, pero son reversibles al descontinuar el medicamento; la atención medica será brindada en el Instituto Nacional de Rehabilitación en el área de Urgencias; usted puede acudir directamente y el medico tratante dará aviso inmediato al coordinador Clínico, Dr Eric Hazan Lasri. El contacto de los médicos responsables se encuentra al final del consentimiento. Además, si usted llegara a ser positivo en los estudios de RT-PCR para SARS-CoV-2 realizados a los 30 o 60 días (es decir, si se confirmara que usted tiene la infección) se valorará individualmente su caso para tomar las medidas e iniciar manejos dictados por la Secretaria de Salud, y quedaría suspendido del resto de la investigación. Si usted llegara a tener complicaciones la atención de las mismas no tendrán ningún costo para usted.
- 15. ¿Qué sucede cuando la investigación termina? Las muestras de sangre se procesarán en el laboratorio del grupo de Investigación del ELEVATE Trial, el laboratorio se encuentra en la Unidad de Medicina Regenerativa en el quinto piso de la torre de Investigación, en las instalaciones del Instituto Nacional de Rehabilitación. Las muestras serán codificadas para garantizar la confidencialidad de datos personales y tan sólo las personas directamente relacionadas con la investigación tendrán acceso a los detalles de las muestras biológicas. Así mismo, el conocimiento adquirido se divulgará en medios científicos y habrá una transferencia de este a otros centros de salud. Las muestras serán almacenadas por lo menos 5 años a partir del fin de la investigación.
- 16. ¿A quién puedo dirigirme si tengo alguna complicación, preocupación o problema relacionado con la Investigación? El responsable, o investigador principal y coordinador de esta investigación, es el Dr. Julio Granados Montiel, teléfono 5554329237, con horario de lungarente.





"2021, Año de la Independencia"

viernes de 7 a 15 hrs, correo electrónico juliogram@gmail.com. También puede comunicarse con el Dr. Eric Hazan Lasri, teléfono 5585814488 extensión 12102, con horario de lunes a viernes de 8 a 15 hrs, correo electrónico doctorhazan@gmail.com, o directamente llamar al servicio de Urgencias del Instituto Nacional de Rehabilitación "Luis Guillermo Ibarra Ibarra", teléfono 555999-1000 extensión 17103 o 17212, en caso de requerir atención inmediata por alguna complicación relacionada con esta investigación. El médico adscrito de guardia estará atendiéndolo.

## **ACLARACIONES**

- a) Esta investigación ha sido revisada y aprobada por el Comité de Investigación y Comité de Ética en Investigación del Instituto Nacional de Rehabilitación "Luis Guillermo Ibarra Ibarra", que son independientes al grupo de investigadores, para proteger sus intereses como participante.
- b) Su decisión de participar en la presente Investigación es completamente voluntaria.
- c) En el transcurso de la Investigación, usted podrá solicitar información actualizada sobre la misma, al investigador responsable.
- d) La información obtenida en esta investigación, utilizada para la identificación de cada participante, será mantenida con estricta confidencialidad, conforme la normatividad vigente.
- e) Se le garantiza que usted recibirá respuesta a cualquier pregunta, duda o aclaración acerca de los procedimientos, riesgos, beneficios u otros asuntos relacionados con la presente investigación.
- f) Se hace de su conocimiento que existe la disponibilidad de tratamiento médico y la indemnización a que legalmente tendría derecho por parte del Instituto Nacional de Rehabilitación "Luis Guillermo Ibarra Ibarra", solamente en el caso de sufrir daños directamente causados por la Investigación.
- g) En caso de que sea usted padre/tutor, o representante legal de un menor de edad o de una persona incapaz de tomar la decisión o firmar este documento, sírvase firmar la presente Carta de Consentimiento Informado dando su autorización.
- h) En el caso de que el participante en la investigación se trate de un menor a partir de los 6 años, por favor de lectura al Asentimiento Informado anexo a este documento, para que el menor lo comprenda y autorice.
- i) Si considera que no hay dudas ni preguntas acerca de su participación, puede, si así lo desea, firmar la Carta de Consentimiento Informado.
- j) Se le comunica que esta Carta de Consentimiento Informado se elabora y firma en dos ejemplares originales, se le entregará un original y el otro lo conservará el investigador principal.







## "2021, Año de la Independencia" FIRMA DE CONSENTIMIENTO [Versión 1, fecha 02/05/2020]

| mi voluntad participar en esta i | nvestigación titulada: "Nuevo<br>de la salud con dosis bajas de | manifiesto que fui ticipación y en pleno uso de mis facultades, es régimen de PROFILAXIS para infección por Hidroxicloroquina y Bromhexina. Un ensayo Trial)". |
|---|---|---|
| | | ampliamente, respecto de los procedimientos ue estaré expuesto ya que dicho procedimiento |
| | | is preguntas han sido respondidas de manera |
| NOMBRE Y FIRMA DEL | | NOMBRE Y FIRMA DEL |
| PARTICIPANTE, PADRE/ | TUTOR O | INVESTIGADOR PRINCIPAL |
| REPRESENTANTE LEGA | L | |
| (según aplique, se requiere ide | entificación) | |
| | TESTIGOS | |
| NOMBRE Y FIRMA | | NOMBRE Y FIRMA |
| PARENTESCO | | PARENTESCO |
| DOMICILIO | | DOMICILIO |

Nota: Los datos personales contenidos en la presente Carta de Consentimiento Informado, serán protegidos conforme a lo dispuesto en las Leyes Federal de Transparencia y Acceso a la Información Pública, General de Transparencia y Acceso a la Información Pública y General de Protección de Datos Personales en Posesión de Sujetos Obligados y demás normatividad aplicable en la materia.

